CLINICAL TRIAL: NCT04517396
Title: FEnofibRate as a Metabolic INtervention for Coronavirus Disease 2019
Brief Title: FEnofibRate as a Metabolic INtervention for COVID-19
Acronym: FERMIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Arizona (Other); Universidad Católica de Santa María (Other); Hospital Nacional Adolfo Guevara Velasco (Other); Hospital Nacional Edgardo Rebagliati Martins (Other); Hospital Nacional Alberto Sabogal Sologuren (Other); Hospital Nacional Guillermo Almenara Irigoyen (Other); Hospital Nacional Carlos Alberto Seguin Escobedo - EsSalud (Other); Universidad de Santander (Other); National Center for Advancing Translational Sciences (NCATS) (NIH); Hospital Civil de Guadalajara (Other); Hospital Nacional Dos De Mayo (Other); Hospital Central Fuerza Aérea del Perú (Other); Hospital Militar Central.Coronel Luis Arias Schereiber (Other); Hospital Victor Lazarte Echegaray (Other); University Hospital, Ioannina (Other); AHEPA University Hospital (Other); Sotiria Thoracic Diseases Hospital of Athens (Other); Thriasio General Hospital of Elefsina (Other); University Hospital, Alexandroupolis (Other); G.Gennimatas General Hospital (Other); Biomelab S.A.S. (Industry); Fundación Oftalmológica de Santander. Santander, Colombia (Other); IPS Centro Científico Asistencial. Barranquilla, Colombia (Other); Fundación Cardiomet. Quindio, Colombia (Other); ClÍnica de Marly (Other); Clínica Internacional (Other)
Responsible Party: Principal Investigator, Julio A. Chirinos, Associate Professor of Medicine at the Hospital of the University of Pennsylvania, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 843729
Record Dates: First submitted 2020-08-17; First posted 2020-08-18 (Actual); Results first posted 2023-02-27 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Fenofibrate; fenofibric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fenofibrate + Usual Care (Experimental): The randomized intervention will be Fenofibrate, in combination with usual care. Dosing: 145 mg of Tricor or a dose-equivalent preparation
  Interventions: Other: Fenofibrate/fenofibric acid; Other: Usual care
- Placebo + Usual Care (Placebo Comparator): The randomized intervention will a matching placebo, in combination with usual care.
  Interventions: Other: Placebo; Other: Usual care

INTERVENTIONS:
Other: Fenofibrate/fenofibric acid — The randomized intervention will be fenofibrate (Tricor) at a dose of 145 mg/d or dose-equivalent preparation of fenofibrate or fenofibric acid, for 10 days. In all cases, appropriate dose reductions will be implemented for patients with chronic kidney disease as per the approved preparation label. The intended duration of randomized treatment will be for 10 days.
  Arms: Fenofibrate + Usual Care
Other: Placebo — The control intervention will be a placebo, for 10 days.
  Arms: Placebo + Usual Care
Other: Usual care — All participants will otherwise receive usual medical care

SUMMARY:
The severe acute respiratory syndrome coronavirus 2 (SARS-CoC-2), the virus responsible for coronavirus disease 2019 (COVID-19), is associated with a high incidence of acute respiratory distress syndrome (ARDS) and death. Aging, obesity, diabetes, hypertension and other risk factors associated with abnormal lipid and carbohydrate metabolism are risk factors for death in COVID-19. Recent studies suggest that COVID-19 progression is dependent on metabolic mechanisms. Moreover, gene expression analyses in cultured human bronchial cells infected with SARS-CoV-2 and lung tissue from patients with COVID-19, indicated a marked shift in cellular metabolism, with excessive intracellular lipid generation. In this cell culture system, fenofibrate (a widely available low-cost generic drug approved by the FDA and multiple other regulatory agencies around the world to treat dyslipemias) at concentrations that can be achieved clinically, markedly inhibited SARS-CoV-2 viral replication. Fenofibrate also has immunomodulatory effects that may be beneficial in the setting of COVID-19. The aim of this trial is to assess the clinical impact of fenofibrate (145 mg/d of Tricor or dose-equivalent preparations for 10 days, with dose adjustment in chronic kidney disease ([CKD]) to improve clinical outcomes in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of COVID-19, based on: (a) A compatible clinical presentation with a positive laboratory test for SARS-CoV-2, or (b) Considered by the primary team to be a Person Under Investigation undergoing testing for COVID-19 with a high clinical probability, in addition to compatible pulmonary infiltrates on chest x-ray (bilateral, intersticial or ground glass opacities) or chest CT.
* Able to provide informed consent.
* Fewer than 14 days since symptom onset.

Exclusion Criteria:

* Known pregnancy or breastfeeding
* Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2 or undergoing dialysis (CKD stages 4-5).
* History of active liver disease, cholelithiasis, uncontrolled hypothyroidism, or rhabdomyolysis (suspected or confirmed). Patients with a history of hypothyroidism receiving a stable dose of thyroid replacement therapy for at least 6 weeks, with a documented normal TSH (primary hypothyroidism) or free thyroxine (secondary or tertiary hypothyroidism) level at least 6 weeks after the last dose change will be considered eligible for enrollment.
* Known hypersensitivity to fenofibrate or fenofibric acid.
* Ongoing treatment with fenofibrate, clofibrate, warfarin and other coumarin anticoagulants, glimepiride, cyclosporine, tacrolimus
* Use of statins other than simvastatin, pravastatin or atorvastatin ≤40 mg/d or rosuvastatin ≤20 mg/d
* Prisoners/incarcerated individuals
* Inability to read, write or no access to a smart phone, computer or tablet device
* Intubated patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Not making it available

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Bornstein SR, Dalan R, Hopkins D, Mingrone G, Boehm BO. Endocrine and metabolic link to coronavirus infection. Nat Rev Endocrinol. 2020 Jun;16(6):297-298. doi: 10.1038/s41574-020-0353-9. PMID 32242089
- [Background] Yang JK, Feng Y, Yuan MY, Yuan SY, Fu HJ, Wu BY, Sun GZ, Yang GR, Zhang XL, Wang L, Xu X, Xu XP, Chan JC. Plasma glucose levels and diabetes are independent predictors for mortality and morbidity in patients with SARS. Diabet Med. 2006 Jun;23(6):623-8. doi: 10.1111/j.1464-5491.2006.01861.x. PMID 16759303
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Wu C, Chen X, Cai Y, Xia J, Zhou X, Xu S, Huang H, Zhang L, Zhou X, Du C, Zhang Y, Song J, Wang S, Chao Y, Yang Z, Xu J, Zhou X, Chen D, Xiong W, Xu L, Zhou F, Jiang J, Bai C, Zheng J, Song Y. Risk Factors Associated With Acute Respiratory Distress Syndrome and Death in Patients With Coronavirus Disease 2019 Pneumonia in Wuhan, China. JAMA Intern Med. 2020 Jul 1;180(7):934-943. doi: 10.1001/jamainternmed.2020.0994. PMID 32167524
- [Background] Zhu L, She ZG, Cheng X, Qin JJ, Zhang XJ, Cai J, Lei F, Wang H, Xie J, Wang W, Li H, Zhang P, Song X, Chen X, Xiang M, Zhang C, Bai L, Xiang D, Chen MM, Liu Y, Yan Y, Liu M, Mao W, Zou J, Liu L, Chen G, Luo P, Xiao B, Zhang C, Zhang Z, Lu Z, Wang J, Lu H, Xia X, Wang D, Liao X, Peng G, Ye P, Yang J, Yuan Y, Huang X, Guo J, Zhang BH, Li H. Association of Blood Glucose Control and Outcomes in Patients with COVID-19 and Pre-existing Type 2 Diabetes. Cell Metab. 2020 Jun 2;31(6):1068-1077.e3. doi: 10.1016/j.cmet.2020.04.021. Epub 2020 May 1. PMID 32369736
- [Background] McBride CE, Machamer CE. Palmitoylation of SARS-CoV S protein is necessary for partitioning into detergent-resistant membranes and cell-cell fusion but not interaction with M protein. Virology. 2010 Sep 15;405(1):139-48. doi: 10.1016/j.virol.2010.05.031. Epub 2010 Jul 1. PMID 20580052
- [Background] Ehrlich E, Uhl S, Ioannidis K, Hofree M, tenOever B, Nahmias Y. The SARS-CoV-2 Transcriptional Metabolic Signature in Lung Epithelium. Cell Sneak Peak (submission only). 2020
- [Background] Schaefer MB, Pose A, Ott J, Hecker M, Behnk A, Schulz R, Weissmann N, Gunther A, Seeger W, Mayer K. Peroxisome proliferator-activated receptor-alpha reduces inflammation and vascular leakage in a murine model of acute lung injury. Eur Respir J. 2008 Nov;32(5):1344-53. doi: 10.1183/09031936.00035808. Epub 2008 Jul 24. PMID 18653653
- [Background] Hecker M, Behnk A, Morty RE, Sommer N, Vadasz I, Herold S, Seeger W, Mayer K. PPAR-alpha activation reduced LPS-induced inflammation in alveolar epithelial cells. Exp Lung Res. 2015;41(7):393-403. doi: 10.3109/01902148.2015.1046200. PMID 26151160
- [Background] Huang D, Zhao Q, Liu H, Guo Y, Xu H. PPAR-alpha Agonist WY-14643 Inhibits LPS-Induced Inflammation in Synovial Fibroblasts via NF-kB Pathway. J Mol Neurosci. 2016 Aug;59(4):544-53. doi: 10.1007/s12031-016-0775-y. Epub 2016 Jun 24. PMID 27339772
- [Background] Ling H, Luoma JT, Hilleman D. A Review of Currently Available Fenofibrate and Fenofibric Acid Formulations. Cardiol Res. 2013 Apr;4(2):47-55. doi: 10.4021/cr270w. Epub 2013 May 9. PMID 28352420
- [Background] Ladabaum U, Mannalithara A, Myer PA, Singh G. Obesity, abdominal obesity, physical activity, and caloric intake in US adults: 1988 to 2010. Am J Med. 2014 Aug;127(8):717-727.e12. doi: 10.1016/j.amjmed.2014.02.026. Epub 2014 Mar 11. PMID 24631411
- [Background] O'Connor CM, Whellan DJ, Fiuzat M, Punjabi NM, Tasissa G, Anstrom KJ, Benjafield AV, Woehrle H, Blase AB, Lindenfeld J, Oldenburg O. Cardiovascular Outcomes With Minute Ventilation-Targeted Adaptive Servo-Ventilation Therapy in Heart Failure: The CAT-HF Trial. J Am Coll Cardiol. 2017 Mar 28;69(12):1577-1587. doi: 10.1016/j.jacc.2017.01.041. PMID 28335841
- [Background] Margulies KB, Hernandez AF, Redfield MM, Givertz MM, Oliveira GH, Cole R, Mann DL, Whellan DJ, Kiernan MS, Felker GM, McNulty SE, Anstrom KJ, Shah MR, Braunwald E, Cappola TP; NHLBI Heart Failure Clinical Research Network. Effects of Liraglutide on Clinical Stability Among Patients With Advanced Heart Failure and Reduced Ejection Fraction: A Randomized Clinical Trial. JAMA. 2016 Aug 2;316(5):500-8. doi: 10.1001/jama.2016.10260. PMID 27483064
- [Background] Felker GM, Maisel AS. A global rank end point for clinical trials in acute heart failure. Circ Heart Fail. 2010 Sep;3(5):643-6. doi: 10.1161/CIRCHEARTFAILURE.109.926030. No abstract available. PMID 20841546
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Hozo SP, Djulbegovic B, Hozo I. Estimating the mean and variance from the median, range, and the size of a sample. BMC Med Res Methodol. 2005 Apr 20;5:13. doi: 10.1186/1471-2288-5-13. PMID 15840177
- [Background] Julious SA. Sample sizes for clinical trials with normal data. Stat Med. 2004 Jun 30;23(12):1921-86. doi: 10.1002/sim.1783. PMID 15195324
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341
- [Background] PASS 16 Power Analysis and Sample Size Software. NCSS, LLC. Kaysville, Utah, USA, ncss.com/software/pass. 2018
- [Background] Fay MP, Malinovsky Y. Confidence intervals of the Mann-Whitney parameter that are compatible with the Wilcoxon-Mann-Whitney test. Stat Med. 2018 Nov 30;37(27):3991-4006. doi: 10.1002/sim.7890. Epub 2018 Jul 8. PMID 29984411
- [Background] Willan AR, Pater JL. Carryover and the two-period crossover clinical trial. Biometrics. 1986 Sep;42(3):593-9. PMID 3567292
- [Background] Brown BW Jr. The crossover experiment for clinical trials. Biometrics. 1980 Mar;36(1):69-79. PMID 7370374
- [Background] GRIZZLE JE. THE TWO-PERIOD CHANGE-OVER DESIGN AN ITS USE IN CLINICAL TRIALS. Biometrics. 1965 Jun;21:467-80. No abstract available. PMID 14338679
- [Background] Therneau TM, Grambsch PM. Modeling Survival Data: Extending the Cox Model. In: Statistics for Biology and Health. New York, NY: Springer; 2001
- [Background] Little RJ. Modeling the drop-out mechanism in repeated-measures studies. Journal of the American Statistical Association. 1995;90:1112-1121
- [Background] Li P, Stuart EA, Allison DB. Multiple Imputation: A Flexible Tool for Handling Missing Data. JAMA. 2015 Nov 10;314(18):1966-7. doi: 10.1001/jama.2015.15281. No abstract available. PMID 26547468
- [Background] Tahmaz M, Kumbasar B, Ergen K, Ure U, Karatemiz G, Kazancioglu R. Acute renal failure secondary to fenofibrate monotherapy-induced rhabdomyolysis. Ren Fail. 2007;29(7):927-30. doi: 10.1080/08860220701573640. PMID 17994463
- [Background] Ghosh B, Sengupta S, Bhattacharjee B, Majumder A, Sarkar SB. Fenofibrate-induced myopathy. Neurol India. 2004 Jun;52(2):268-9. PMID 15269493
- [Background] Zhou J, Li D, Cheng Q. Fenofibrate monotherapy-induced rhabdomyolysis in a patient with post-pancreatitis diabetes mellitus: A rare case report and a review of the literature. Medicine (Baltimore). 2020 May 22;99(21):e20390. doi: 10.1097/MD.0000000000020390. PMID 32481339
- [Background] Keech A, Simes RJ, Barter P, Best J, Scott R, Taskinen MR, Forder P, Pillai A, Davis T, Glasziou P, Drury P, Kesaniemi YA, Sullivan D, Hunt D, Colman P, d'Emden M, Whiting M, Ehnholm C, Laakso M; FIELD study investigators. Effects of long-term fenofibrate therapy on cardiovascular events in 9795 people with type 2 diabetes mellitus (the FIELD study): randomised controlled trial. Lancet. 2005 Nov 26;366(9500):1849-61. doi: 10.1016/S0140-6736(05)67667-2. PMID 16310551
- [Background] Davidson MH. Reducing residual risk for patients on statin therapy: the potential role of combination therapy. Am J Cardiol. 2005 Nov 7;96(9A):3K-13K; discussion 34K-35K. doi: 10.1016/j.amjcard.2005.08.002. Epub 2005 Sep 12. PMID 16291008
- [Background] Guo J, Meng F, Ma N, Li C, Ding Z, Wang H, Hou R, Qin Y. Meta-analysis of safety of the coadministration of statin with fenofibrate in patients with combined hyperlipidemia. Am J Cardiol. 2012 Nov 1;110(9):1296-301. doi: 10.1016/j.amjcard.2012.06.050. Epub 2012 Jul 27. PMID 22840347
- [Background] Davidson MH, Rooney MW, Drucker J, Eugene Griffin H, Oosman S, Beckert M; LCP-AtorFen Investigators. Efficacy and tolerability of atorvastatin/fenofibrate fixed-dose combination tablet compared with atorvastatin and fenofibrate monotherapies in patients with dyslipidemia: a 12-week, multicenter, double-blind, randomized, parallel-group study. Clin Ther. 2009 Dec;31(12):2824-38. doi: 10.1016/j.clinthera.2009.12.007. PMID 20110022
- [Background] ACCORD Study Group; Ginsberg HN, Elam MB, Lovato LC, Crouse JR 3rd, Leiter LA, Linz P, Friedewald WT, Buse JB, Gerstein HC, Probstfield J, Grimm RH, Ismail-Beigi F, Bigger JT, Goff DC Jr, Cushman WC, Simons-Morton DG, Byington RP. Effects of combination lipid therapy in type 2 diabetes mellitus. N Engl J Med. 2010 Apr 29;362(17):1563-74. doi: 10.1056/NEJMoa1001282. Epub 2010 Mar 14. PMID 20228404
- [Background] Bergman AJ, Murphy G, Burke J, Zhao JJ, Valesky R, Liu L, Lasseter KC, He W, Prueksaritanont T, Qiu Y, Hartford A, Vega JM, Paolini JF. Simvastatin does not have a clinically significant pharmacokinetic interaction with fenofibrate in humans. J Clin Pharmacol. 2004 Sep;44(9):1054-62. doi: 10.1177/0091270004268044. PMID 15317833
- [Background] Whitfield LR, Porcari AR, Alvey C, Abel R, Bullen W, Hartman D. Effect of gemfibrozil and fenofibrate on the pharmacokinetics of atorvastatin. J Clin Pharmacol. 2011 Mar;51(3):378-88. doi: 10.1177/0091270010366446. Epub 2010 Apr 22. PMID 20413454
- [Background] Patino-Rodriguez O, Martinez-Medina RM, Torres-Roque I, Martinez-Delgado M, Mares-Garcia AS, Escobedo-Moratilla A, Covarrubias-Pinedo A, Arzola-Paniagua A, Herrera-Torres JL, Perez-Urizar J. Absence of a significant pharmacokinetic interaction between atorvastatin and fenofibrate: a randomized, crossover, study of a fixed-dose formulation in healthy Mexican subjects. Front Pharmacol. 2015 Jan 29;6:4. doi: 10.3389/fphar.2015.00004. eCollection 2015. PMID 25688207
- [Background] Backman JT, Kyrklund C, Kivisto KT, Wang JS, Neuvonen PJ. Plasma concentrations of active simvastatin acid are increased by gemfibrozil. Clin Pharmacol Ther. 2000 Aug;68(2):122-9. doi: 10.1067/mcp.2000.108507. PMID 10976543
- [Background] Kyrklund C, Backman JT, Neuvonen M, Neuvonen PJ. Gemfibrozil increases plasma pravastatin concentrations and reduces pravastatin renal clearance. Clin Pharmacol Ther. 2003 Jun;73(6):538-44. doi: 10.1016/S0009-9236(03)00052-3. PMID 12811363
- [Background] Schneck DW, Birmingham BK, Zalikowski JA, Mitchell PD, Wang Y, Martin PD, Lasseter KC, Brown CD, Windass AS, Raza A. The effect of gemfibrozil on the pharmacokinetics of rosuvastatin. Clin Pharmacol Ther. 2004 May;75(5):455-63. doi: 10.1016/j.clpt.2003.12.014. PMID 15116058
- [Background] Guiomar V, Oliveira D, Correia C, Pereira E. Efficacy of Rituximab in Refractory Inflammatory Myopathy Associated With Coexistence of Behcet's Disease and Antiphospholipid Syndrome. Eur J Case Rep Intern Med. 2019 Nov 11;6(11):001294. doi: 10.12890/2019_001294. eCollection 2019. PMID 31890711
- [Background] Atmaca H, Sayarlioglu H, Kulah E, Demircan N, Akpolat T. Rhabdomyolysis associated with gemfibrozil-colchicine therapy. Ann Pharmacother. 2002 Nov;36(11):1719-21. doi: 10.1345/aph.1C028. PMID 12398566
- [Background] Sugie M, Kuriki A, Arai D, Ichikawa H, Kawamura M. [A case report of acute neuromyopathy induced by concomitant use of colchicine and bezafibrate]. No To Shinkei. 2005 Sep;57(9):785-90. Japanese. PMID 16248366
- [Background] Feher MD, Hepburn AL, Hogarth MB, Ball SG, Kaye SA. Fenofibrate enhances urate reduction in men treated with allopurinol for hyperuricaemia and gout. Rheumatology (Oxford). 2003 Feb;42(2):321-5. doi: 10.1093/rheumatology/keg103. PMID 12595630
- [Background] Schlesinger N. Management of acute and chronic gouty arthritis: present state-of-the-art. Drugs. 2004;64(21):2399-416. doi: 10.2165/00003495-200464210-00003. PMID 15481999
- [Background] Lee YH, Lee CH, Lee J. Effect of fenofibrate in combination with urate lowering agents in patients with gout. Korean J Intern Med. 2006 Jun;21(2):89-93. doi: 10.3904/kjim.2006.21.2.89. PMID 16913436
- [Background] Jung JY, Choi Y, Suh CH, Yoon D, Kim HA. Effect of fenofibrate on uric acid level in patients with gout. Sci Rep. 2018 Nov 13;8(1):16767. doi: 10.1038/s41598-018-35175-z. PMID 30425304
- [Background] Khanna PP. Gout: a patrician malady no more. Lancet Diabetes Endocrinol. 2018 Apr;6(4):263-264. doi: 10.1016/S2213-8587(18)30073-1. No abstract available. PMID 29571506
- [Background] Waldman B, Ansquer JC, Sullivan DR, Jenkins AJ, McGill N, Buizen L, Davis TME, Best JD, Li L, Feher MD, Foucher C, Kesaniemi YA, Flack J, d'Emden MC, Scott RS, Hedley J, Gebski V, Keech AC; FIELD investigators. Effect of fenofibrate on uric acid and gout in type 2 diabetes: a post-hoc analysis of the randomised, controlled FIELD study. Lancet Diabetes Endocrinol. 2018 Apr;6(4):310-318. doi: 10.1016/S2213-8587(18)30029-9. Epub 2018 Feb 26. PMID 29496472
- [Background] Ting R-D, Keech A. Fenofibrate and renal disease: clinical effects in diabetes. Clinical Lipidology. 2013;8(6):669-680
- [Background] McDonald KB, Garber BG, Perreault MM. Pancreatitis associated with simvastatin plus fenofibrate. Ann Pharmacother. 2002 Feb;36(2):275-9. doi: 10.1345/aph.1A180. PMID 11847949
- [Background] Enger C, Gately R, Ming EE, Niemcryk SJ, Williams L, McAfee AT. Pharmacoepidemiology safety study of fibrate and statin concomitant therapy. Am J Cardiol. 2010 Dec 1;106(11):1594-601. doi: 10.1016/j.amjcard.2010.07.041. Epub 2010 Oct 14. PMID 21094360
- [Derived] Chirinos JA, Lopez-Jaramillo P, Giamarellos-Bourboulis EJ, Davila-Del-Carpio GH, Bizri AR, Andrade-Villanueva JF, Salman O, Cure-Cure C, Rosado-Santander NR, Cornejo Giraldo MP, Gonzalez-Hernandez LA, Moghnieh R, Angeliki R, Cruz Saldarriaga ME, Pariona M, Medina C, Dimitroulis I, Vlachopoulos C, Gutierrez C, Rodriguez-Mori JE, Gomez-Laiton E, Cotrina Pereyra R, Ravelo Hernandez JL, Arbanil H, Accini-Mendoza J, Perez-Mayorga M, Milionis C, Poulakou G, Sanchez G, Valdivia-Vega R, Villavicencio-Carranza M, Ayala-Garcia RJ, Castro-Callirgos CA, Alfaro Carrasco RM, Garrido Lecca Danos W, Sharkoski T, Greene K, Pourmussa B, Greczylo C, Ortega-Legaspi J, Jacoby D, Chittams J, Katsaounou P, Alexiou Z, Sympardi S, Sweitzer NK, Putt M, Cohen JB; FERMIN Investigators. A randomized clinical trial of lipid metabolism modulation with fenofibrate for acute coronavirus disease 2019. Nat Metab. 2022 Dec;4(12):1847-1857. doi: 10.1038/s42255-022-00698-3. Epub 2022 Nov 7. PMID 36344766
- [Derived] Chirinos J, Lopez-Jaramillo P, Giamarellos-Bourboulis E, Davila-Del-Carpio G, Bizri A, Andrade-Villanueva J, Salman O, Cure-Cure C, Rosado-Santander N, Giraldo MC, Gonzalez-Hernandez L, Moghnieh R, Angeliki R, Saldarriaga MC, Pariona M, Medina C, Dimitroulis I, Vlachopoulos C, Gutierrez C, Rodriguez-Mori J, Gomez-Laiton E, Pereyra R, Hernandez JR, Arbanil H, Accini-Mendoza J, Perez-Mayorga M, Milionis H, Poulakou G, Sanchez G, Valdivia-Vega R, Villavicencio-Carranza M, Ayala-Garcia R, Castro-Callirgos C, Carrasco RA, Danos WL, Sharkoski T, Greene K, Pourmussa B, Greczylo C, Chittams J, Katsaounou P, Alexiou Z, Sympardi S, Sweitzer N, Putt M, Cohen J. A Randomized Trial of Lipid Metabolism Modulation with Fenofibrate for Acute Coronavirus Disease 2019. Res Sq [Preprint]. 2022 Aug 10:rs.3.rs-1933913. doi: 10.21203/rs.3.rs-1933913/v1. PMID 35982675

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fenofibrate + Usual Care | Placebo + Usual Care
Started | 351 | 350
Completed | 347 | 347
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fenofibrate + Usual Care | Placebo + Usual Care | Total
Number analyzed (Participants) | 351 | 350 | 701
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 293 | 289 | 582
  >=65 years | 58 | 61 | 119
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 166 | 330
  Male | 187 | 184 | 371
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 173 | 177 | 350
  Not Hispanic or Latino | 178 | 173 | 351
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 24 | 25 | 49
  White | 168 | 170 | 338
  More than one race | 133 | 134 | 267
  Unknown or Not Reported | 21 | 20 | 41
Region of Enrollment [Number; unit: participants]
  United States | 57 | 59 | 116
  Mexico | 34 | 33 | 67
  Peru | 58 | 58 | 116
  Colombia | 79 | 77 | 156
  Greece | 67 | 66 | 133
  Lebanon | 56 | 57 | 113
Borg Scale [Mean (Standard Deviation); unit: units on a scale] — This is a scale that asks participants to rate the difficulty of their breathing. The scale starts at number 0 where breathing is causing no difficulty at all and progresses through to number 10 where breathing difficulty is maximal. The total Borg scale is reported. Please see the following reference for additional information: https://www.cdc.gov/physicalactivity/basics/measuring/exertion.htm
  units on a scale | 2.6 (2.8) | 2.9 (3.1) | 2.7 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Primary Hierarchical Composite Endpoint
Description: The primary endpoint of the trial is a global rank score that ranks patient outcomes according to 5 factors. The global rank score, or global severity score, is a nonparametric, hierarchically ranked outcome. The global rank score was generated by ranking all 701 participants on a scale of 1 to 701, from worst to best clinical outcomes. Participants were ranked by (1) time to death; (2) the number of days supported by invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); (3) The inspired concentration of oxygen/percent oxygen saturation (FiO2/SpO2) ratio area under the curve; (4) For participants enrolled as outpatients who are subsequently hospitalized, the number of days out of the hospital during the 30 day-period following randomization; (5) For participants enrolled as outpatients who don't get hospitalized during the 30-day observation period, the modified Borg dyspnea scale
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: Ranked Severity Score
Arm/Group | Fenofibrate + Usual Care | Placebo + Usual Care
Number analyzed (Participants) | 351 | 350
Ranked Severity Score | 5.32 [2.98 to 6.00] | 5.33 [2.98 to 6.00]

2. Secondary Outcome: Number of Days Alive, Out of the Intensive Care Unit, Free of Mechanical Ventilation/Extracorporeal Membrane Oxygenation, or Maximal Available Respiratory Support in the 30 Days Following Randomization
Description: Number of days participants were alive, out of the intensive care unit, free of mechanical ventilation/extracorporeal membrane oxygenation, or maximal available respiratory support during the 30 days that followed randomization
Time Frame: Up to 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Fenofibrate + Usual Care | Placebo + Usual Care
Number analyzed (Participants) | 351 | 350
days | 28.8 (4.9) | 28.3 (6.1)

3. Secondary Outcome: Seven-category Ordinal Scale
Description: A seven-category ordinal scale consisting of the following categories: 1, not hospitalized with resumption of normal activities; 2, not hospitalized, but unable to resume normal activities; 3, hospitalized, not requiring supplemental oxygen; 4, hospitalized, requiring supplemental oxygen; 5, hospitalized, requiring nasal high-flow oxygen therapy, noninvasive mechanical ventilation, or both; 6, hospitalized, requiring extracorporeal membrane oxygenation (ECMO), invasive mechanical ventilation, or both; and 7, death.
Time Frame: At 15 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fenofibrate + Usual Care | Placebo + Usual Care
Number analyzed (Participants) | 351 | 350
score on a scale | 1 [1 to 1] | 1 [1 to 2]

4. Secondary Outcome: Secondary Hierarchical Composite Endpoint
Description: The secondary global rank score, or global severity score, is a nonparametric, hierarchically ranked outcome. The global rank score was generated by ranking all 701 participants on a scale of 1 to 701, from worst to best clinical outcomes. Participants were ranked by (1) time to death; (2) the number of days supported by invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); (3) The inspired concentration of oxygen/percent oxygen saturation (FiO2/SpO2) ratio area under the curve; (4) For participants enrolled as outpatients who are subsequently hospitalized, the number of days out of the hospital during the 30 day-period following randomization; (5) For participants enrolled as outpatients who don't get hospitalized during the 30-day observation period, a COVID-19 symptom scale rating fever, cough, dyspnea, muscle aches, sore throat, loss of smell or taste, headache, diarrhea, fatigue, nausea/vomiting, chest pain (each are rated from 0-10 then summed).
Time Frame: Up to 30 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fenofibrate + Usual Care | Placebo + Usual Care
Number analyzed (Participants) | 351 | 350
score on a scale | 5.05 [2.98 to 5.22] | 5.05 [2.98 to 5.21]

5. Other Pre Specified Outcome: All-Cause Death
Description: Death from any cause during the observation period
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Fenofibrate + Usual Care | Placebo + Usual Care
Number analyzed (Participants) | 351 | 350
Participants | 19 | 22

6. Other Pre Specified Outcome: Number of Days Alive and Out of the Hospital During the 30 Days Following Randomization
Description: Number of days that participants were alive and out of the hospital during the 30 days following randomization
Time Frame: Up to 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fenofibrate + Usual Care | Placebo + Usual Care
Number analyzed (Participants) | 351 | 350
days | 30 [25 to 30] | 30 [25 to 30]

7. Other Pre Specified Outcome: Exploratory Hierarchical Composite Endpoint
Description: The exploratory global rank score, or global severity score, is a nonparametric, hierarchically ranked outcome. The global rank score was generated by ranking all 701 participants on a scale of 1 to 701, from worst to best clinical outcomes. Participants were ranked by (1) time to death; (2) the number of days supported by invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); (3) The inspired concentration of oxygen/percent oxygen saturation (FiO2/SpO2) ratio area under the curve; (4) The number of days out of the hospital during the 30 day-period following randomization.
Time Frame: Up to 30 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fenofibrate + Usual Care | Placebo + Usual Care
Number analyzed (Participants) | 351 | 350
score on a scale | 5.03 [2.98 to 5.03] | 5.03 [2.98 to 5.03]

ADVERSE EVENTS:
Time Frame: 30 days post-randomization
Description: The research team kept a log of all adverse events in the trial. A medically-qualified investigator assessed all AEs, which were classified by organ system category.
  The definition of adverse events and Serious Adverse Events (SAE) is presented in detail in the study protocol, available in this clinicaltrials.gov record (protocol sections 4.1, 4.2 and 4.3)
Arm/Group | Fenofibrate + Usual Care | Placebo + Usual Care
All-Cause Mortality (participants affected / at risk) | 19/351 | 22/350
Serious Adverse Events (participants affected / at risk) | 46/351 | 61/350
Other Adverse Events (participants affected / at risk) | 74/351 | 55/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenofibrate + Usual Care (N=351) | Placebo + Usual Care (N=350)
Intensive Care Unit Transfer (General disorders) | 13 (13) | 16 (17)
Death (General disorders) | 19 (19) | 22 (22)
Invasive mechanical ventilation (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 16 (16)
Acute Coronary Syndrome (Cardiac disorders) | 9 (10) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 3 (3)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
New or worsening cognitive status (Psychiatric disorders) | 5 (5) | 2 (2)
Liver failure or acute liver injury (Hepatobiliary disorders) | 2 (2) | 9 (11)
Acute kidney injury (Renal and urinary disorders) | 7 (16) | 12 (14)
Suspected or confirmed rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Worsening dyspnea or hypoxia (Respiratory, thoracic and mediastinal disorders) | 23 (23) | 31 (32)
Superimposed infection (Infections and infestations) | 7 (8) | 4 (4)
New or worsening diarrhea, nausea, or vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Other new or worsening neurologic issues (Nervous system disorders) | 2 (2) | 2 (2)
Other (General disorders) | 11 (18) | 16 (21)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenofibrate + Usual Care (N=351) | Placebo + Usual Care (N=350)
Kidney (Renal and urinary disorders) | 8 (11) | 10 (19)
Hepatic (Hepatobiliary disorders) | 20 (25) | 16 (24)
Cardiovascular (Cardiac disorders) | 8 (8) | 8 (10)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 5 (10)
Gastroenterologic (Gastrointestinal disorders) | 16 (17) | 5 (5)
Infectious (Infections and infestations) | 24 (45) | 21 (30)
Neurologic (Nervous system disorders) | 3 (5) | 3 (3)
Dermatologic (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Endocrinologic (Endocrine disorders) | 1 (1) | 2 (2)
Hematologic (Blood and lymphatic system disorders) | 9 (12) | 10 (13)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Other (General disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
The study enrolled participants over an 18-month period where several different SARS-CoV-2 variants dominated, and national interventions and vaccine availability varied at different timepoints. Additionally, components of the hierarchical endpoints may be subjective.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/96/NCT04517396/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-06): https://cdn.clinicaltrials.gov/large-docs/96/NCT04517396/SAP_001.pdf